CLINICAL TRIAL: NCT03053648
Title: Self-acupressure for Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Self-acupressure for Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEAR 20161123005
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Insomnia; Acupressure
Keywords: Insomnia; Randomized controlled trial; Acupressure; Self-help
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All of the assessments in this study will be self-completed. The researchers who perform the assessment and analysis will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-acupressure Group (Experimental): Subjects in this group will attend two weekly 120-minute self-acupressure training sessions in a classroom at the School of Nursing, the Hong Kong Polytechnic University. The subjects will be instructed on how to perform the self-acupressure treatment by a trained instructor. To enhance interaction and ensure the quality of teaching, each course will be conducted in a small group of 6 participants. Subjects will perform self-acupressure daily for 4 consecutive weeks.
  Interventions: Other: Self-acupressure
- Sleep Hygiene Education Group (Active Comparator): To control the contact time with professional person in the treatment group, participants in this group will receive two sessions of 120-minute sleep hygiene training session. The participants will be asked to follow the health hygiene instructions daily for 4 consecutive weeks.
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Other: Self-acupressure — The subjects will be told to perform self-acupressure 30 min before sleep for 20 min every night for 4 weeks. Telephone follow-up will be made twice a week by the trained student research assistant during the 4-week treatment period to remind subjects to practice self-acupressure.
  Arms: Self-acupressure Group
Other: Sleep hygiene education — A training hand-out will be provided to each subject. The hand-outs included manualized sleep hygiene instructions. A registered nurse who has been trained by a clinical psychologist will be the instructor on sleep hygiene and activity scheduling. To enhance interaction and ensure the quality of teaching, each course will be conducted in a group of 5 participants.
  Arms: Sleep Hygiene Education Group

SUMMARY:
Abstract

Objectives: To explore the clinical effects of self-acupressure for treating insomnia delivered by a training course.

Hypothesis: Subjects who have participated in the self-acupressure training course will have greater improvement in insomnia symptoms and daytime impairment than the sleep hygiene education control group at 4 and 8 weeks.

Design and subjects: A pilot randomized controlled trial. Subjects with insomnia will be recruited from the community. 30 subjects will be randomized to self-acupressure and sleep hygiene education control groups in a 1: 1 ratio. Study instrument: Insomnia Severity Index (ISI) will be used to assess insomnia symptoms and daytime impairment.

Interventions: Subjects in the self-acupressure group will attend two training sessions to learn self-acupressure and will practice self-acupressure every night for 4 weeks; subjects in the sleep hygiene education control group will receive two training sessions to learn sleep hygiene practice.

Main outcome measures: The primary outcome measure is the ISI score. Other measures include sleep parameters using subjective sleep diary, Hospital Anxiety and Depression Scale, and SF-6D at 4 and 8 weeks. Acceptability and sustainability of self-acupressure will also be evaluated.

Data Analysis: Differences in the questionnaire scores, subjective sleep parameters will be examined using a mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

* (1) Chinese Hong Kong residents who are able to communicate in Cantonese or Putonghua;
* (2) Aged 18 - 65 years;
* (3) A current clinical Diagnostic and Statistical Manual of Mental Disorders, Fifth edition (DSM-5) diagnosis of insomnia disorder according to the Brief Insomnia Questionnaire (BIQ), a validated diagnostic tool. (The criteria include having difficulties in falling asleep, difficulties in staying asleep, or early morning awakening with clinically significant consequences for daily life for at least 3 months.)
* (4) Insomnia Severity Index total score of at least 10 indicating insomnia at the clinical level; and
* (5) Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

* (1) Receiving acupuncture or practitioner-delivered acupressure treatment in the past 6 months;
* (2) Pregnancy;
* (3) Cognitive impairment as indicated by a Mini Mental State Examination ≤ 23;
* (4) At significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (score ≥ 3);
* (5) No comorbid sleep disorders primarily requiring other treatment, such as sleep apnea or narcolepsy; and
* (6) Taking herbal remedies, over-the-counter medication, or psychotropic drugs that target insomnia within the 2 weeks prior to baseline.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-03 (Estimated); Study Completion 2017-03-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 7 days
  The ISI is a seven-item self-rating scale. The subjects rate the severity of insomnia, the distress, and the functional impairment associated with insomnia on a 5-point Likert scale.

SECONDARY OUTCOMES:
The 7-day daily sleep diary | 7 days
  The standardized sleep diary records the bedtime and rising time, from which the total time in bed (TIB) can be calculated. Subjects will be asked to estimate sleep-onset latency, wake after sleep onset, and total sleep time (TST). Sleep efficiency will be calculated as (TST/TIB * 100%).
Hospital Anxiety and Depression Scale (HADS) | 7 days
  The HADS is a 14-item self-administrated questionnaire, which assess the severity of depressive and anxiety symptoms.
Short Form-6D (SF-6D) | 4 weeks
  SF-6D is composed of six multi-level dimensions: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality.

CONTACTS AND LOCATIONS:
Overall Officials: Wing-Fai Yeung, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong